CLINICAL TRIAL: NCT06804707
Title: Tissue and Vascular Microstructure Evaluation for Carotid Plaque Characterization Using Innovative Ultrasound Techniques
Brief Title: Carotid Plaque Characterization Using Innovative Ultrasound Techniques
Acronym: CARPUS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL24_0689
Record Dates: First submitted 2025-01-27; First posted 2025-02-03 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-01

CONDITIONS: Carotid Atheroma
Keywords: Carotid atheroma; Plaque characterization; Ultrasound; Ultrasound Localization Microscopy; Backscatter Coefficient; Vasa vasorum; Intraplaque Hemorrhage
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: This is a single-center, cross-sectional, descriptive and exploratory study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- patients with carotid plaque (Experimental): Patients over 18 years of age with asymptomatic or symptomatic carotid plaque with a degree of stenosis > 50% North American Symptomatic Carotid Endarterectomy Trial (NASCET) from vascular surgery consultations and for whom a surgical indication has been retained
  Interventions: Biological: blood sampling; Device: ultrasound imaging exam; Device: High resolution MRI plaque exam

INTERVENTIONS:
Biological: blood sampling — This procedure will take place once during the patient's CARPUS first visit (Croix Rousse hospital (Hospice civils de Lyon).
  A peripheral venous line of the cathlon 24 G type with tap without tubing will be inserted by a nurse. A blood sample will be taken at the same time to check creatinine levels before the MRI scan and to record the patient's cholesterol levels for the eCRF.
Device: ultrasound imaging exam — This procedure takes place once immediately after the intervention 1. The patient will first have an ultrasound acquisition with the clinical ultrasound scanner (~5 minutes) in order to locate the plaque. An acquisition with the research ultrasound scanner and matrix probe will then be performed for measurement for ultrasound spectroscopy (~5 minutes).
  An injection of 2.4 ml Sonovue followed by 10 ml saline will be performed during acquisition with the research ultrasound scanner for ultrasound localization imaging measurement (~10 minutes).
  The patient must remain under observation (in the waiting room) for 30 minutes after the examination.
Device: High resolution MRI plaque exam — This procedure will take place once during the patient's CARPUS second visit (Pierre Wertheimer hospital (Hospice civils de Lyon)).
  The patient is greeted in radiology, and his/her identity and absence of contraindications are verified.
  A peripheral venous line of the cathlon 24 G type with tap without tubing will be inserted by a nurse.
  Injection of gadolinium and MRI examination of the plaque used in clinical routine.

SUMMARY:
Strokes are the second leading cause of disability and death worldwide (according to World Health Organization in 2019). They are ischemic in origin in 80% of cases. Atheromatous disease, and more specifically carotid stenosis, is responsible for 20% of these ischemic strokes. Current recommendations, based on high levels of evidence, consider only the degree of carotid artery stenosis to define the threshold for surgical treatment. However, it is now accepted that the composition and rate of progression of atherosclerotic plaque are also criteria to be considered when selecting patients at high risk of stroke. The presence of hemorrhage and a lipid core in the atheromatous plaque, both factors of instability, is associated with a greater risk of ipsilateral ischemic events. The presence of intraplaque hemorrhage is therefore a marker of plaque instability. In this context, techniques for in vivo analysis of atherosclerotic plaque composition need to be developed to better target patients for surgery.

Ultrafast ultrasound enables imaging rates of several thousand images per second. Ultrasound Localization Microscopy (ULM) gives access to the vascular microstructure of tissues: the localization of injected microbubbles, which enhance the ultrasound signal in vessels, and the tracking of these microbubbles enable the vascularization of the tissue in question to be mapped. Ultrasound spectroscopy qualifies tissue microstructure: this operator- and system-independent technique is based on frequency analysis of ultrasound signals backscattered by tissue, and more specifically on analysis of the backscatter coefficient (BSC). Measuring the BSC is intrinsic to the tissue, and provides quantitative parameters on the scatterers to qualify the tissue.

The study hypothesis is that these two ultrasound techniques will provide information on the characteristics of the atherosclerotic plaque: the presence of neovessels and biomarkers linked to its composition, including intraplaque hemorrhage.

ELIGIBILITY:
Inclusion Criteria:

* Female or male over 18 years of age
* Patients with asymptomatic or symptomatic carotid plaque (stenosis> 50% NASCET), referred by the Hospices Civils de Lyon (HCL) vascular surgery consultation and for whom a surgical indication has been retained.
* Patient having agreed to participate in the study and signed a written informed consent form
* Patient affiliated to a social security scheme or equivalent.

Exclusion Criteria:

* Patients with contraindications to Sonovue (right-to-left shunt, severe pulmonary hypertension, allergy to the molecule)
* Patients with unstable cardiovascular pathology (coronary artery disease, stroke / transient ischemic attack, cardiac rhythm disorders)
* Uncontrolled hypertension
* Respiratory distress syndrome
* Patients with contraindications to MRI (claustrophobia, presence of metallic elements, etc.).
* Gadolinium-related contraindications and precautions for use
* Contraindication to dobutamine
* Hypersensitivity to the active substance or to one of the constituents of Gadolinium,
* Renal insufficiency with clearance <30 ml/min/1.73 m²,
* Pregnant or breast-feeding patients
* Patients under guardianship or trusteeship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2025-03-10 (Estimated); Primary Completion 2027-01-10 (Estimated); Study Completion 2027-01-10 (Estimated)

PRIMARY OUTCOMES:
Volume of neovessels in carotid atherosclerotic plaques by ULM | between 6 and 59 days after inclusion
  From the vascularization cartography obtained by ULM, the volume of vascularization of the plaque will be estimated (number of pixels with vascularization compared with the number of pixels in the plaque x100). Plaques can then be described by neovessel volume distribution.
Mean velocity in neovessels in carotid atherosclerotic plaques by ULM | between 6 and 59 days after inclusion
  From the vascularization cartography obtained by ULM, the mean velocity (mm/s) in all the neovessels will be estimated.
Location of neovessels in carotid atherosclerotic plaques by ULM | between 6 and 59 days after inclusion
  The main location of vessels will also be described according to their topography in the plaque (e.g. central, peripheral, both).

SECONDARY OUTCOMES:
Lizzi Feleppa slope (dB/MHz) derived from BSC measured by ultrasound spectroscopy on carotid atherosclerotic plaques | between 6 and 59 days after inclusion
  In ultrasound signals, the plaque is divided into regions of interest and ultrasound spectroscopy is applied. This will enable us to obtain the backscatter coefficient (BSC) for each region of interest. From the backscatter coefficient, parameters derived from the BSC will be evaluated.
  One of these parameters is:
  - Lizzi-Feleppa slope: slope of the linear fit of the BSC as a function of frequency.
  This parameter in the different regions of interest on the plaque will be averaged for each plaque.
Lizzi Feleppa intercept (dB) derived from BSC measured by ultrasound spectroscopy on carotid atherosclerotic plaques | between 6 and 59 days after inclusion
  In ultrasound signals, the plaque is divided into regions of interest and ultrasound spectroscopy is applied. This will enable us to obtain the backscatter coefficient (BSC) for each region of interest. From the backscatter coefficient, parameters derived from the BSC will be evaluated.
  One of these parameters is:
  - Lizzi-Feleppa intercept: intercept of the linear fit of the BSC as a function of frequency.
  This parameter in the different regions of interest on the plaque will be averaged for each plaque.
Lizzi Feleppa midband (dB) derived from BSC measured by ultrasound spectroscopy on carotid atherosclerotic plaques | between 6 and 59 days after inclusion
  In ultrasound signals, the plaque is divided into regions of interest and ultrasound spectroscopy is applied. This will enable us to obtain the backscatter coefficient (BSC) for each region of interest. From the backscatter coefficient, parameters derived from the BSC will be evaluated.
  One of these parameters is:
  - Lizzi-Feleppa midband: midband of the linear fit of the BSC as a function of frequency.
  This parameter in the different regions of interest on the plaque will be averaged for each plaque.
Integrated backscatter coefficient (BSC) (dB) measured by ultrasound spectroscopy on carotid atherosclerotic plaques | between 6 and 59 days after inclusion
  In ultrasound signals, the plaque is divided into regions of interest and ultrasound spectroscopy is applied. This will enable us to obtain the backscatter coefficient (BSC) for each region of interest. From the backscatter coefficient, parameters derived from the BSC will be evaluated.
  One of these parameters is:
  - integrated BSC: Integrated BSC on the -6 dB frequency bandwidth.
  This parameter in the different regions of interest on the plaque will be averaged for each plaque.
Acoustic attenuation (dB/mm) measured by ultrasound on carotid atherosclerotic plaques | between 6 and 59 days after inclusion
  In ultrasound signals, the plaque is divided into regions of interest and ultrasound spectroscopy is applied. This will enable us to obtain the backscatter coefficient (BSC) for each region of interest. From the backscatter coefficient, parameters derived from the BSC will be evaluated.
  One of these parameters is:
  - acoustic attenuation.
  This parameter in the different regions of interest on the plaque will be averaged for each plaque.
Correlation between the volume of neovessels in carotid atherosclerotic plaques, estimated by ULM, and that estimated by anatomopathological analyses | between 6 and 59 days after inclusion
  For each plaque, histological analysis will give the stage of intraplaque haemorrhage according to Derksen's grading scale if intraplaque haemorrhage is present. A semi-quantitative grading denoting the quantity of neovessels (score between 0 and 3) will also be performed. The correlation between these grades and the volume of neovessels originating from the ULM will be studied.
Correlation between ultrasound parameters of BSC related to intraplaque hemorrhage of carotid atherosclerotic plaques and intraplaque hemorrhage assessed by anatomopathological analyses | between 6 and 59 days after inclusion
  Histological analysis will give the stage of intraplaque haemorrhage according to Derksen's grading scale if intraplaque haemorrhage is present. A semi-quantitative scale denoting the ratio of the area of intraplaque hemorrhage to the total area of the plaque (score 0 if ratio between 0 and 25%, score 1 if ratio between 25 and 50%, score 2 if ratio between 50 and 75% and score 3 if ratio between 75 and 100%). The thresholds for the BSC parameters need to be calibrated to determine the thresholds corresponding to intraplaque hemorrhage. For this step, areas of intraplaque hemorrhage will be localized using plaque MRI. This will enable us to determine which BSC parameter or combination of parameters best characterizes intraplaque hemorrhage, and then to estimate for each plaque a relative volume of region of interest containing intraplaque hemorrhage.
  The correlation between these grades and the volume of intraplaque hemorrhage derived from ultrasound measurements will be studied.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Ariane BLEROT, MD, PhD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital de la Croix Rousse, Lyon, France

IPD SHARING:
Plan to Share IPD: No